CLINICAL TRIAL: NCT03497767
Title: A Randomised Phase II Trial of Osimertinib With or Without Stereotactic Radiosurgery for EGFR Mutated Non-Small Cell Lung Cancer (NSCLC) With Brain Metastases
Brief Title: A Randomised Phase II Trial of Osimertinib With or Without SRS for EGFR Mutated NSCLC With Brain Metastases
Acronym: OUTRUN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 17.02
Record Dates: First submitted 2018-02-26; First posted 2018-04-13 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer (NSCLC); EGFR mutation; Osimertinib; Stereotactic Radiosurgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osimertinib (Experimental): 80mg Osimerinib taken once daily
  Interventions: Drug: Osimertinib
- Stereotactic Radiosurgery + Osimertinib (Experimental): Upfront Stereotactic Radiosurgery (SRS) followed by 80mg Osimerinib taken once daily
  Interventions: Drug: Osimertinib; Radiation: Stereotactic Radiosurgery (SRS)

INTERVENTIONS:
Drug: Osimertinib — All participants will receive a dose of Osimertinib 80mg once daily
  Other Names: Tagrisso
Radiation: Stereotactic Radiosurgery (SRS) — Dose and fractionation depend on lesion size. All SRS must be completed within 21 days of randomisation and all lesions are to be treated within 7 days.
  Arms: Stereotactic Radiosurgery + Osimertinib

SUMMARY:
20-40% of patients with NSCLC will develop brain metastases at some point during their course of disease. Osimertinib has demonstrated intracranial activity in EFGR mutated NSCLC with leptomeningeal disease in the phase 1 BLOOM study. Stereotactic radiosurgery (SRS) is one of the standard local treatment for patients with limited number of brain metastases. Currently, it is unclear whether adding SRS to Osimertinib will result in superior intracranial disease control in patients with EGFR mutated NSCLC with brain metastases diagnosed de novo or developed while on first line EGFR tyrosine kinase inhibitors (TKIs) such as Erlotinib and Gefinitib.

The aim of this study is to compare the effects of Osimertinib alone versus SRS plus Osimertinib on intra-cranial disease control in EGFR mutated NSCLC with brain metastases diagnosed or developed while on first line EGFR tyrosine kinase inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent
2. Has reached the age of majority in the country of treatment (i.e. ≥ 18 years in Australia; ≥ 21 years in Singapore)
3. Histological or cytological documented NSCLC
4. Metastatic NSCLC, not amenable to curative surgery or curative radiotherapy
5. Brain metastases that meet the following criteria;

   1. ≤ 10 lesion/s visible and measurable on protocol screening MRI;

      * At least one brain metastases able to be treated with SRS
      * Definite but small brain metastases not for SRS treatment due to size, as per physician discretion, are included in the total
      * Equivocal small lesions are not included in the total
   2. No single brain metastasis exceeding 30mm longest diameter
   3. Total brain metastasis volume ≤ 15cc;

      - Total brain metastases volume on protocol screening MRI should be using the formula (4/3) x (3.14159265359) x (1/2 x size lesion in centimetre)3. Table 1: Brain metastases volume estimates provides an estimate of the volume of brain metastases based on the size of the lesion
   4. Diagnosed de novo (i.e. at the same time with a new diagnosis of NSCLC) or developed as a new site of progression while on first line EGFR TKI

   NOTE: Surgery as part of local practice for the management of brain metastasis is allowed but must be completed between 2 to 4 weeks prior to randomisation. Patients must still fulfil criteria 5a, 5b and 5d pre-surgery, and have at least one target lesion post-surgery to be eligible for the study. Lesions that are partially or completely resected should not be used as a target lesion for MRI assessment.
6. Documented EGFR mutation;

   1. Patients who developed brain metastases as a site of disease progression while on first line EGFR TKIs must have T790M mutation.
   2. Documented EGFR mutation (at any time since the initial diagnosis of NSCLC) known to be sensitive to Osimertinib - These include exon 19 del; L858R (exon 21); G719X (exon 18); L861G (exon 21); S768I (exon 20) and T790M (exon 20) NOTE: Mutation analysis is to be done as per local practice. Please see section 7.1.1 for the recommended clinical practice for analysis.
7. Are one of the following cohorts:

   1. First-line metastatic cancer: All newly diagnosed participants with documented sensitising EGFR mutation (criterion 6) and intracranial metastasis (criterion 5), with/without extracranial disease
   2. Second-line metastatic cancer (T790M+): Participants who progressed after first-line 1st or 2nd generation EGFR TKI therapy with intracranial progression (criterion 5), with/without extracranial disease and have documented T790M mutation
   3. Second-line metastatic cancer (T790M-): Participants with no T790M mutation who progressed after first-line 1st or 2nd generation EGFR TKI therapy with intracranial progression (criterion 5) but has no extracranial disease
   4. Second-line metastatic cancer (T790M-): Participants with no T790M mutation who progressed after first-line 1st or 2nd generation EGFR TKI therapy with intracranial progression (criterion 5) but has stable extracranial disease
8. Karnofsky performance status 60-100 (ECOG performance status ≤2) with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks
9. Female patients who;

   1. are willing to use adequate contraceptive measures until 6 weeks after the final dose of study treatment
   2. are not breast feeding
   3. have a negative pregnancy test prior to the start of dosing if of child bearing potential or have evidence of non-child bearing potential by fulfilling one of the following criteria at screening:

   i. Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments ii. Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with Luteinizing Hormone (LH) and Follicle-Stimulating Hormone (FSH) levels in the post-menopausal range for the institution iii. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
10. Male patients who are willing to use barrier contraception (i.e. condoms) until 4 months after the final dose of study treatment

Exclusion criteria:

1. Treatment with any of the following:

   1. Prior systemic therapy for patients with newly diagnosed metastatic NSCLC and brain metastases de novo.

      NOTE: Prior adjuvant chemotherapy or chemotherapy used as radio sensitisation followed by maintenance immunotherapy for non-resectable early stage NSCLC are allowed if such treatments were more than 6 months ago.
   2. Prior whole brain radiotherapy (WBRT)
   3. Radiologically progressive brain metastasis that underwent prior SRS (second line patients)
   4. Previous treatment with Osimertinib or a 3rd generation EGFR TKI.
   5. Previous treatment with checkpoint inhibitors immunotherapy for metastatic NSCLC.
   6. Major surgery within 4 weeks of randomisation (excluding placement of vascular access and surgery as part of local practice for the management of brain metastases, as outlined in inclusion criterion 5).
   7. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of randomisation.
   8. Medications or herbal supplements known to be potent inducers of CYP3A4 and are unable to stop use within the recommended wash out period prior to receiving the first dose of Osimertinib, see Table 7: Medications to avoid and withdrawal periods and Table 8 NOTE: All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4
   9. An investigational drug within five half-lives of the compound or 3 months, whichever is greater.
   10. Any other cytotoxic chemotherapy, investigational agents or other anticancer drugs from a previous treatment regimen or clinical study within 14 days of randomisation.
2. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 (with the exception of alopecia grade 2) at the time of starting study treatment.
3. Spinal cord compression unless asymptomatic and stable.
4. Leptomeningeal disease.
5. Moderate or severe symptomatic brain metastases defined as per Radiation Therapy Oncology Group acute morbidity grade 3 to 4.

   NOTE:
   * Grade 3 refers to neurological findings requiring hospitalisation for initial management.
   * Grade 4 refers to serious neurological impairment including paralysis, coma or seizures more than three times per week despite medication and requires hospitalization.
6. Brain metastases in the brainstem.
7. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
8. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of Osimertinib.
9. Any of the following cardiac criteria:

   1. Resting corrected QT interval (QTc) > 470 msec, obtained from an electrocardiogram (ECG).
   2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block or second degree heart block.
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including: Serum/plasma potassium < LLN; Serum/plasma magnesium < LLN; Serum/plasma calcium < LLN), congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
10. Patients with congenital long QT syndrome (CLQTS)
11. Past medical history of Interstitial Lung Disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
12. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

    1. Absolute neutrophil count < 1.5 X 109/L
    2. Platelet count < 100 X 109/L
    3. Haemoglobin < 90 g/L
    4. Alanine aminotransferase (ALT) > 2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases
    5. Aspartate aminotransferase (AST) > 2.5 times ULN if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases.
    6. Total bilirubin > 1.5 times ULN if no liver metastases or > 3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases.
    7. Creatinine > 1.5 times ULN concurrent with creatinine clearance < 50ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is > 1.5 times ULN.
13. History of hypersensitivity of drugs with a similar chemical structure or class to Osimertinib or any excipients of these agents.
14. Involvement in the planning and conduct of the study
15. Judgement by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Intracranial progression free survival at 12 months | 12 months post randomisation
  To assess the efficacy of Osimertinib with deferred local brain metastases directed therapies compared with upfront SRS followed by Osimertinib by assessment of intracranial progression free survival at 12 months.

SECONDARY OUTCOMES:
Use of salvage whole-brain radiotherapy (WBRT) | 18 months post randomisation
  To assess the effect of Osimertinib with deferred local brain metastases directed therapies compared with upfront SRS followed by Osimertinib on use of salvage whole-brain radiotherapy (WBRT) +/- neurosurgery.
Local brain failure | 18 months post randomisation
  To assess the effect of Osimertinib with deferred local brain metastases directed therapies compared with upfront SRS followed by Osimertinib on local brain failure.
Distant brain failure | 18 months post randomisation
  To assess the effect of Osimertinib with deferred local brain metastases directed therapies compared with upfront SRS followed by Osimertinib on distant brain failure.
Extra-cranial progression | 18 months post randomisation
  To assess the effect of Osimertinib with deferred local brain metastases directed therapies compared with upfront SRS followed by Osimertinib on extra-cranial progression.
Overall Survival | 18 months post randomisation
  To further assess the efficacy of Osimertinib with deferred local brain metastases directed therapies compared with upfront SRS followed by Osimertinib in terms of overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Hegi-Johnson, Dr, Study Chair — Peter MacCallum Cancer Centre, Australia; Chee Lee, Dr, Study Chair — National Health and Medical Research Council, Australia; Ivan Tham, Dr, Study Chair — National University Hospital, Singapore; Yu Yang Soon, Dr, Study Chair — National University Hospital, Singapore
Locations (13):
- Australia (12):
  - Calvary Mater, Newcastle, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - St. Vincents Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Blacktown Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - ICON Cancer Centre Greenslopes, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Center, Melbourne, Victoria
  - Monash Health, Melbourne, Victoria
  - Sir Charles Gairdner, Perth, Western Australia
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee CK, Lefresne S, Soon YY, Robledo K, Nichol A, Sahgal A, Pinkham MB, Melosky B, Huang Y, McDermott R, Tham IWK, Parmar A, Tey JCS, Liu M, Solomon BJ, Sacher A, Leong CN, Laskin J, Koh WY, Menjak IB, Ang Y, Shultz DB, Low JL, Doherty M, Yong C, Lim MC, Tan AP, Soo RA, Hegi-Johnson F, Ho C. Osimertinib and Stereotactic Radiosurgery for Brain Metastases in EGFR-Mutated Lung Cancer: The STARLET Joint Analysis of OUTRUN and LUOSICNS Randomized Trials. J Thorac Oncol. 2026 Jan 12:103549. doi: 10.1016/j.jtho.2026.01.001. Online ahead of print. PMID 41534788
- See also: Sponsor's webpage — https://trog.com.au/trials/trog-17-02-outrun/